CLINICAL TRIAL: NCT06973889
Title: Evaluation of IgY Antibodies Effectiveness in Egg Yolk Against Helicobacter Pylori in Removing Bacteria and Improving Clinical Symptoms in the Patients
Brief Title: Evaluation of IgY Antibody Efficacy in Egg Yolk Against Helicobacter Pylori in Bacterial Elimination and Clinical Symptoms Improvement of Gastrointestinal Patients
Acronym: Hp IgY
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Mashhad University of Medical Sciences (Other)
Responsible Party: Principal Investigator, zahra esmaeili, Student, Mashhad University of Medical Sciences
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: IR.MUMS.REC.1401.381
Record Dates: First submitted 2025-05-07; First posted 2025-05-15 (Actual); Last update posted 2025-05-15 (Actual); Status verified 2025-05

CONDITIONS: HELICOBACTER PYLORI INFECTIONS; Gastrointestinal Disease
Keywords: IgY; Helicobacter pylori; clinical trial; Antibody; gastrointestinal disease
MeSH Terms: conditions — Gastrointestinal Diseases

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Intervention (Experimental): 12 grams of egg yolk powder containing about 2 grams of antibody twice a day for 2 weeks along with usual antibiotic treatment including OAC or omeprazole (40 mg/day), clarithromycin (1000 mg/day) and amoxicillin (2000 mg/day).
  Interventions: Biological: Helicobacter pylori eradication therapy
- Control (No Intervention): normal egg yolk powder without IgY in the amount of 12 grams 2 times a day for 2 weeks along with usual antibiotic treatment OAC or omeprazole (40 mg/day), clarithromycin (1000 mg/day) and amoxicillin (2000 mg/day)

INTERVENTIONS:
Biological: Helicobacter pylori eradication therapy — 12 grams of egg yolk powder containing about 2 grams of antibody twice a day for 2 weeks along with usual antibiotic treatment including OAC or omeprazole (40 mg/day), clarithromycin (1000 mg/day) and amoxicillin (2000 mg/day).
  Arms: Intervention

SUMMARY:
1. Investigating its effectiveness in removing bacteria in invivo conditions
2. Investigating the effectiveness in improving the clinical symptoms of patients

ELIGIBILITY:
Inclusion Criteria:

* Patients with gastritis or stomach ulcers whose Helicobacter infection has been confirmed by a doctor and age group 18 to 78 years, all genders, if accepted

Exclusion Criteria:

* Acute perforation of esophagus, stomach and duodenum Hyperlipidemic people Those who are allergic to egg proteins Patients with stomach cancer

Ages: 18 Years to 78 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Actual)
Dates: Start 2023-12-04 (Actual); Primary Completion 2024-12-30 (Actual); Study Completion 2025-01-21 (Actual)

PRIMARY OUTCOMES:
Respiratory urea level (UBT) higher than cut off 50 | Determination of respiratory urea (UBT) at the beginning of the study and 8 weeks after the start of the intervention
  This test is performed with the help of a diagnostic kit. After oral ingestion of a capsule containing labeled carbon and the patient's exhalation into the kit, the amount of urea breathed in is determined by the device. A UBT value greater than 50 means Helicobacter pylori infection.

SECONDARY OUTCOMES:
Examining the patient's clinical symptoms including: abdominal pain, nausea, vomiting and bloating. | During the treatment period for 4 weeks from the beginning of the intervention.
  Based on the scoring of gastrointestinal symptoms (GSRS) in such a way that the score is calculated as follows: the number of participants with reduced abdominal pain: 0 (no symptoms), 1 (mild means the presence of tolerable symptoms), 2 (moderate means discomfort and interference) in normal activities), 3 (severe means inability to perform normal activities) -- the number of participants with reduced gastrointestinal symptoms: 0 (absence of nausea), 1 (temporary and short periods of nausea), 2 (frequent nausea) and long-term without vomiting), 3 (persistent nausea and frequent vomiting) -- the number of participants with reduced bloating: 0 (no bloating), 1 (short-term and temporary bloating), 2 (long-term but tolerable bloating), 3 (severe flatulence and interference in social functioning)

CONTACTS AND LOCATIONS:
Locations (2):
- Iran (2):
  - Mashhad University of Medical Sciences, Mashhad, Khorasan
  - Mashhad university of medical sciences, Mashhad, Khorasan

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Suzuki H, Nomura S, Masaoka T, Goshima H, Kamata N, Kodama Y, Ishii H, Kitajima M, Nomoto K, Hibi T. Effect of dietary anti-Helicobacter pylori-urease immunoglobulin Y on Helicobacter pylori infection. Aliment Pharmacol Ther. 2004 Jul;20 Suppl 1:185-92. doi: 10.1111/j.1365-2036.2004.02027.x. PMID 15298626